CLINICAL TRIAL: NCT01856699
Title: Observational Study on the Prognostic Relevance of Supratentorial Superficial Siderosis in Patients With Suspected Cerebral Amyloid Angiopathy
Brief Title: Superficial Siderosis in Patients With Suspected Cerebral Amyloid Angiopathy
Acronym: SuSPect-CAA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Christian Opherk, Principal Investigator, Ludwig-Maximilians - University of Munich
Other Study IDs: SuSPect-CAA
Record Dates: First submitted 2013-05-15; First posted 2013-05-17 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Intracerebral Hemorrhage; Cerebral Amyloid Angiopathy; Ischemic Stroke
Keywords: supratentorial superficial siderosis; intracerebral hemorrhage; cerebral amyloid angiopathy
MeSH Terms: conditions — Cerebral Hemorrhage; Cerebral Amyloid Angiopathy; Ischemic Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, plasma, CSF
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study Group: Patients with cortical superficial siderosis and possible or probable cerebral amyloid angiopathy meeting the modified Boston criteria.
- Control Group: Patients with possible or probable cerebral amyloid angiopathy meeting the classic Boston criteria but without any cortical superficial siderosis.

SUMMARY:
Aim of the SuSPect-CAA study is to prospectively evaluate the prognostic significance of cortical superficial siderosis in patients with suspected cerebral amyloid angiopathy with a primary focus on future stroke and mortality.

DETAILED DESCRIPTION:
Non-traumatic cortical superficial siderosis (cSS) is a common finding in patients with cerebral amyloid angiopathy (CAA) and can be its sole imaging sign. The clinical features and course as well as the prognostic significance of cSS in CAA patients remain unclear. In a retrospective study we have previously shown that cSS might be an important predictor or warning sign for future intracranial hemorrhage. However, prospective data are missing.

The Superficial Siderosis in Patients with suspected Cerebral Amyloid Angiopathy (SuSPect-CAA) study is designed as a prospective observational multi-centre cohort study. Primary objective of the study is to evaluate if cSS is a predictor for future stroke and mortality (primary endpoint: combined rate of stroke and death after 36 months). Secondary objectives of the study include 1) to evaluate if cSS represents a marker of future intracranial haemorrhage, especially at the site of initial siderosis, 2) to describe the clinical presentation and course of cSS, 3) to assess to associated imaging findings, 4) to determine the differential diagnoses of cSS.

All subjects presenting to the respective neurological centers (out- or inpatient treatment with neuroimaging) will be screened. The study population will consist of two patient groups: 1) Patients meeting the modified Boston criteria for probable or possible CAA, i. e. patients with SS +/- lobar intracerebral hemorrhage or microbleeds in cortico-subcortical localization and absence of other cause of hemorrhage than CAA will be assigned to the study group. 2) Patients meeting the classic Boston criteria for possible or probable CAA but without any SS will be assigned to the control group. A total of 100 patients per group will be enrolled. Baseline and follow-up assessment at 6, 12, 24, and 36 months will be performed by visits in the respective neurological outpatient clinic including a structured interview and neurological exam, neuropsychological tests, EEG and MRI.

ELIGIBILITY:
Inclusion Criteria (study group):

* Fulfillment of the modified Boston criteria for CAA-related hemorrhage with evidence of supratentorial superficial siderosis on MRI
* MR-/CT-/digital subtraction (DS) -angiography without evidence of cerebral aneurysm, arterio-venous malformation (AVM) , AV-fistula or other pathology of relevance (e.g. tumor, hemorrhagic infarction)
* A maximum of two lobar or cerebellar intracranial hemorrhages (ICH) (old or acute)
* Written informed consent by patient or guardian prior to study participation
* Willingness to participate in follow-up

Inclusion Criteria (control group):

* Fulfillment of the classic Boston criteria for CAA-related hemorrhage
* Absence of superficial siderosis on MRI
* A maximum of two lobar or cerebellar ICHs (old or acute)
* MR-/CT-/DS -angiography without evidence of cerebral aneurysm, AVM, AV-fistula or other pathology of relevance (e.g. tumor, hemorrhagic infarction)
* Written informed consent by patient or guardian prior to study participation
* Willingness to participate in follow-up

Exclusion Criteria (both groups):

* Severe medical condition with expected life expectancy <3 years
* More than two lobar or cerebellar ICH (old or acute)
* any intracerebral hemorrhage in the deep grey matter (basal ganglia or thalami) or in the brain stem
* History of head trauma resulting in loss of consciousness or radiologically visible traumatic brain injury (contusions, diffuse axonal damage) in the last 5 years prior to inclusion
* Cerebral aneurysm or history of aneurysmal subarachnoid hemorrhage
* Infratentorial siderosis
* Infratentorial subarachnoid hemorrhage

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospital based
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 2013-05; Primary Completion 2018-12 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Combined rate of stroke and death | 36 months
  All cause mortality and stroke (WHO-definition)

SECONDARY OUTCOMES:
Rate of intracranial hemorrhage | 6, 12, 24, 36 months
  Rate of any intracranial hemorrhage as assessed by cerebral imaging

OTHER OUTCOMES:
Clinical presentation and course of superficial siderosis | 0, 6, 12, 24, 36 months
  A detailed analysis on the clinical presentation and course of superficial siderosis will be performed (detailed questionnaire, comprehensive neurological examinations, disability scales, neuropsychological tests)
Imaging findings associated with superficial siderosis | 0, 6, 12, 24, 36 months
  Localization, extent and progression of superficial siderosis will be assessed on MR-imaging. In addition, the prevalence, incidence, localization, number or extent of cerebral microbleeds, white matter disease, and acute ischemic lesions will be determined using follow-up MRI.
Differential causes of superficial siderosis | 0, 6, 12, 24, 36 months
  At the time of patient screening and follow-up we will systematically evaluate the underlying causes of superficial siderosis and potential differential diagnoses based on the available clinical, laboratory and imaging data, as well as published diagnostic criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Wollenweber, MD, Principal Investigator — Institute for Stroke and Dementia Research, Ludwig-Maximilans-University; Jennifer Linn, MD, Principal Investigator — Department of Neuroradiology, Carl Carus University Dresden; Christian Opherk, MD, Principal Investigator — Institute for Stroke and Dementia Research, Ludwig-Maximilans-University; Martin Dichgans, MD, Study Director — Institute for Stroke and Dementia Research, Ludwig-Maximilians-University
Locations (1):
- Ludwig-Maximilians-University, Munich, Germany

IPD SHARING:
Plan to Share IPD: Undecided